CLINICAL TRIAL: NCT01012804
Title: Assessment of Variation of PKA and Other Molecular Markers in Patients Undergoing Resection of Colon Cancer Metastases
Brief Title: Study of Biomarkers in Tissue Samples From Patients With Metastatic Colon Cancer
Status: Withdrawn | Type: Observational
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: John Marshall, MD, Georgetown University
Other Study IDs: CDR0000078662; P30CA051008 (NIH); GUMC-00074; NCI-G01-1992
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; recurrent colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Blotting, Western; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: western blotting
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This research study is looking at biomarkers in tissue samples from patients with metastatic colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of surgical resection, in terms of physiological stress, on levels of tumor markers such as protein kinase A (PKA) expression in patients with metastatic colon cancer.
* Estimate variation among patients of baseline tumor markers in tumor tissue and sera.
* Correlate markers in tumor tissues with that in sera in these patients.
* Establish a tissue bank of these specimens for future studies.

OUTLINE: Biopsy and surgical specimens are obtained before and during standard surgery (patients may have had tumor tissue obtained before study entry and stored). Serum samples and tumor tissue are analyzed by immunohistochemistry and western blot. Tumor markers (such as PKA expression) are determined and marker levels are measured in serum samples and tissues.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colon cancer

  * Metastatic disease for which surgical resection is indicated
  * Metastatic disease accessible for tissue biopsy OR previously biopsied tissue is available

PATIENT CHARACTERISTICS:

* Platelet count ≥ 80,000/mm^3
* INR ≤ 1.3
* PTT ≤ upper limit of normal
* No history of bleeding disorders or abnormal clotting factors
* No extrahepatic biliary obstruction

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2000-01

CONTACTS AND LOCATIONS:
Overall Officials: John L. Marshall, MD, Study Chair — Lombardi Comprehensive Cancer Center
Locations (1):
- Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia, United States